CLINICAL TRIAL: NCT03917420
Title: Quantification of Estradiol's Impact on Nucleotides in Different Cellular Populations of the Lower Gastrointestinal Tract
Brief Title: Quantification of Estradiol's Impact on Nucleotides in Cellular Populations of the Lower GI Tract
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-0333; R21AI145646 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-04-17 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2019-11

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Tenofovir; Tablets; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tenofovir/Emtricitabine (Experimental): Participants will take 5 once daily doses above noted combination tab at 200mg/300mg before each sampling visit
  Interventions: Drug: Tenofovir 300Mg Oral Tablet; Drug: Emtricitabine 200 MG

INTERVENTIONS:
Drug: Tenofovir 300Mg Oral Tablet — Once daily dose of the combo tab x 5 days pre-sampling
  Other Names: Truvada
Drug: Emtricitabine 200 MG — Once daily dose of the combo tab x 5 days pre-sampling
  Other Names: Truvada

SUMMARY:
Purpose: To Assess the impact of high and low in vivo estradiol exposure on PrEP (Pre-exposure prophylaxis) nucleotide concentrations in different cellular populations of the lower GI (gastrointestinal) tract and to quantify the relationship between estradiol, progesterone, and testosterone on PrEP nucleotide concentrations in rectal and peripheral blood mononuclear cells. As well as the relationship between estradiol, progesterone, and testosterone on PrEP concentrations in plasma.

Participants: Healthy, cisgender female, volunteers, aged 18-49 inclusive on the date of screening with an intact gastrointestinal system and regular menstrual cycle.

Procedures (methods): Participants will take a single daily dose of study drug for five days before each sampling visit. The visits will be scheduled during the early follicular phase of the menstrual cycle (approximately days 2-5 after the first day of menses, Visit 1) when estradiol is predicted to be the lowest and the late follicular phase (approximately days 12-15 after the first day of menses, Visit 2) when estradiol is predicted to be highest. Samples of blood, rectal cells, and rectal tissue will be collected at both Visits 1 and 2. All participants will complete a follow-up safety visit within 14 days of completing study sampling.

DETAILED DESCRIPTION:
Participants will be enrolled, and sampling visits will be scheduled to correspond with their menstrual cycles. Five days prior to the first scheduled sampling visit, participants will come to the clinic to have a repeat urine pregnancy test performed to verify eligibility. After verification, participants will be given a single dose of the study medication, Truvada®. Study staff will witness the dose and assess for any adverse reactions post dose. Participants will be sent home with a supply of 4 additional doses of Truvada® for them to take at scheduled times for the next 4 days with study staff observing via video call. Study staff will assess for adverse events during each dosing call. Starting 72 hours before each sampling visit, participants will be required to switch to a low fiber diet and abstain from inserting anything rectally. Twelve hours prior to each sampling visit, participants will be required to abide by a clear liquid diet. Participants will be seen as an outpatient at the Clinical Translational Research Center (CTRC) at University of North Carolina at Chapel Hill (UNC) for these sampling visits. At these visits, participants will have blood samples drawn to measure peripheral blood mononuclear cells and serum hormone concentrations. Participants will also have rectal cells collected via cytobrush and rectal tissue collected via rectal biopsy. After all samples have been collected, participants will be evaluated for adverse events and be discharged. Within 14 days of completion of the second sampling visit, for a follow-up visit. At this visit, blood will be obtained to check safety labs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy cisgender pre-menopausal female participants between the ages of 18 and 49 years, inclusive on the date of screening (Healthy is defined as no irregular menstrual cycles or clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, and clinical laboratory tests.
* Regular menstrual cycles defined as at least 1 day of menses occurring every 21-35 days)
* Estimated calculated creatinine clearance (eCcr) of at least 60 mL/min by the Cockcroft-Gault formula where: eCcr (female) in mL/min = [(140 - age in years) x (weight in kg) x 0.85] / (72x serum creatinine in mg/dL).
* Negative serum pregnancy test at screening
* All participants should be using at least one of the following methods of contraception* from the screening visit through 72 hours prior to inpatient admission (at which time the women will be asked to remain abstinent until after their follow-up visit):

  1. Non continuous systemic hormonal contraceptives that permit intermittent menstruation
  2. IUD (non-hormonal intrauterine device) placed at least 1 month prior to study enrollment
  3. Bilateral tubal ligation (Sterilization)
  4. Vasectomized male partners
  5. Condom + Spermicide
  6. *Unless engaged in sexual activity with female only sex partners or abstinent for at least 3 months prior with no intention of becoming sexually active during the study period. Any history of recent or present concomitant male sex partners will be addressed and ruled out in the context of screening participants for eligibility for the protocol
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
* Subject must be willing to abstain from sexual intercourse, and all and intrarectal objects and products for at least 72 hours prior to Sampling #1 until study completion.
* Subject must be HIV-1 and Hepatitis B and C negative as documented on screening labs.
* Subject must not be actively involved in the conception process and must be non-lactating.
* Subject must be able to swallow pills and have no allergies to any component of the study product

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including documented drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Participants with a history of hysterectomy
* Participants who are pregnant, possibly pregnant or lactating
* History of febrile illness within five days prior to first dose.
* Any condition possibly affecting drug absorption (eg, gastrectomy or other significant alterations of the gastrointestinal tract)
* A positive urine drug screen.
* An untreated-positive test for syphilis, gonorrhea, or Chlamydia at screening.
* Any clinically relevant laboratory chemistry or hematology result Grade 2 or greater according to the Division of AIDS Laboratory Grading Tables
* Treatment with an investigational drug within 4 months preceding the first dose of study product.
* History of regular alcohol consumption exceeding 14 drinks (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of spirits) per week.
* Participation in a clinical trial involving rectal biopsies within 6 months preceding the first dose of trial medication.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
* Any condition which, in the opinion of the investigator, is likely to interfere with follow-up or ability to take the study medication appropriately.
* Unwilling or unable to comply with the dietary and concomitant drug restrictions in regard to study drug administration as outlined in the study procedures and prohibited medications sections.
* Women utilizing continuous hormonal contraception options such as Seasonique, injectables, implants, and hormonal IUDs

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only cisgender pre-menopausal females will be eligible to enroll
Enrollment: 10 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie Cottrell, PharmD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Response to individual request for raw data. Any resulting publication from this proposal will include the principle investigator or a co-investigator listed on the application as corresponding author. Raw de-identified datasets will be shared with requesting scientists at the discretion of principle investigator to foster scientific openness in an ethical and responsible manner.
Supporting Information: CSR
Time Frame: Upon acceptance of final manuscript for publication for an indefinite time period
Access Criteria: Before data will be shared, a data use agreement will be put in place in accordance with local regulations. The requestor will need to obtain appropriate ethics approval.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tenofovir/Emtricitabine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [20.75 to 30.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Average Tenofovir Diphosphate Concentrations in Mixed Rectal Cells During the Early (Low Estradiol) Follicular Phases of the Menstrual Cycle.
Description: Average tenofovir diphosphate concentrations measured in mixed rectal cells collected via cytobrush during the early (low estradiol) follicular phases of the menstrual cycle reported in Fmol/million cells.
Time Frame: Days 2-5
Measure: Mean (Standard Deviation); unit: fmol/million cells
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
fmol/million cells | 406.14 (819.0428)
Statistical Analysis 1: Comparison: Tenofovir/Emtricitabine; Test type: Other — Correlation; Spearman's Rho = -0.455

2. Primary Outcome: Average Tenofovir Diphosphate Concentrations Measured in Mixed Rectal Cells During the Late (High Estradiol) Follicular Phases of the Menstrual Cycle.
Description: Average tenofovir diphosphate concentrations measured in mixed rectal cells collected via cytobrush during the late (high estradiol) follicular phases of the menstrual cycle reported in Fmol/million cells
Time Frame: Days 12-15
Measure: Mean (Standard Deviation); unit: fmol/million cells
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
fmol/million cells | 480.4 (577.9748)
Statistical Analysis 1: Comparison: Tenofovir/Emtricitabine; Test type: Other — Correlation; Spearman's Rho = 0.152

3. Primary Outcome: Average Emtricitabine Triphosphate Concentrations Measured in Mixed Rectal Cells During the Early (Low Estradiol) Follicular Phases of the Menstrual Cycle.
Description: Average emtricitabine triphosphate concentrations measured in mixed rectal cells collected via cytobrush during the early (low estradiol) follicular phases of the menstrual cycle reported in Fmol/million cells.
Time Frame: Days 2-5
Measure: Mean (Standard Deviation); unit: fmol/million cells
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
fmol/million cells | 13.005 (7.715)
Statistical Analysis 1: Comparison: Tenofovir/Emtricitabine; Test type: Other — Correlation; Spearman's Rho = 0.564

4. Primary Outcome: Average Emtricitabine Triphosphate Concentrations Measured in Mixed Rectal Cells During the Late (High Estradiol) Follicular Phases of the Menstrual Cycle.
Description: Average emtricitabine triphosphate concentrations measured in mixed rectal cells collected via cytobrush during the late (high estradiol) follicular phases of the menstrual cycle reported in Fmol/million cells.
Time Frame: Days 12-15
Measure: Mean (Standard Deviation); unit: fmol/million cells
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
fmol/million cells | 74.822 (97.280)
Statistical Analysis 1: Comparison: Tenofovir/Emtricitabine; Test type: Other — Correlation; Spearman's Rho = 0.285

5. Secondary Outcome: Average Estradiol Concentrations in Serum.
Description: Average estradiol concentrations in serum reported in pg/mL
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
pg/ml | 101.06 (74.52)

6. Secondary Outcome: Average Progesterone Concentrations in Serum.
Description: Average progesterone concentrations in serum measured in ng/mL.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
ng/ml | 2.46 (4.54)

7. Secondary Outcome: Average Testosterone Concentrations in Serum.
Description: Average testosterone concentrations in serum measured in ng/mL
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
ng/ml | 55.45 (21.58)

8. Secondary Outcome: Average Tenofovir Diphosphate Concentrations in Peripheral Blood Mononuclear Cells.
Description: Average tenofovir diphosphate concentrations in peripheral blood mononuclear cells reported in Fmol/million cells.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: Fmol/million cells
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
Fmol/million cells | 96.40 (45.01)

9. Secondary Outcome: Average Emtricitabine Concentrations in Peripheral Blood Mononuclear Cells.
Description: Average emtricitabine concentrations in peripheral blood mononuclear cells reported in Fmol/million cells.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: Fmol/million cells
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
Fmol/million cells | 5601.95 (2235.02)

10. Secondary Outcome: Average Tenofovir Concentrations in Plasma.
Description: Average tenofovir concentrations in plasma reported in ng/mL.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
ng/ml | 61.02 (10.90)

11. Secondary Outcome: Average Emtricitabine Concentrations in Plasma.
Description: Average emtricitabine concentrations in plasma reported in ng/mL.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Tenofovir/Emtricitabine
Number analyzed (Participants) | 10
ng/ml | 78.07 (27.72)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during the interval from study enrollment to follow-up visit, up to a total of 28 days.
Arm/Group | Tenofovir/Emtricitabine
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir/Emtricitabine (N=10)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Viral Pharyngitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT03917420/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT03917420/ICF_001.pdf